CLINICAL TRIAL: NCT02682576
Title: Brachial Artery Ultrasound Imaging: A Repeatability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Everist Genomics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A-1601
Record Dates: First submitted 2016-02-09; First posted 2016-02-15 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Cardiovascular Diseases
Keywords: brachial artery ultrasound imaging; flow-mediated dilation; endothelium
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brachial artery ultrasound imaging (Experimental): Brachial artery ultrasound imaging is a non-invasive procedure for detecting endothelial dysfunction by measuring the flow-mediated dilation of the brachial artery using high resolution continuous electrocardiogram-gated B-mode (2D) ultrasound imaging during reactive hyperemia.
  Interventions: Procedure: Brachial artery ultrasound imaging

INTERVENTIONS:
Procedure: Brachial artery ultrasound imaging

SUMMARY:
The objective of the study is to define the analytical repeatability of quantifying flow-mediated dilation of the brachial artery using brachial artery ultrasound imaging using upper arm cuff occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ≥18 years old
2. Eastern Cooperative Oncology Group/Zubrod score performance status of 0, 1, or 2, determined within 7 days prior to FMD testing on Study Day 1 (Visit 1)
3. Written informed consent understood and signed; understanding of study procedures and ability to comply with them for the length of the study

Exclusion Criteria:

1. Body mass index (BMI) >50 kg/m2
2. Mid-upper arm circumference of arm selected for FMD testing <17 cm or >42 cm
3. Sinus arrhythmia (RR intervals vary by >50%), atrial fibrillation, atrial flutter, multifocal atrial tachycardia, frequent (>1 per 10-sec strip) premature atrial or ventricular contractions (isolated, non-isolated, or alternating), documented by 12-lead ECG with rhythm strip at the time of subject screening.
4. Clinical signs and/or symptoms of active viral or bacterial infections
5. Resting tremor or inability to remain still for the duration of the testing period
6. Systolic blood pressure (SBP) at rest of >170 mmHg or diastolic blood pressure (DBP) at rest of ≥110 mmHg.
7. Diabetic subjects - Type I or II
8. Previous intolerable adverse reaction(s) to vascular testing using an upper extremity occlusive pneumatic cuff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline % flow-mediated dilation (%FMD) at 1 hour | 1 hour
  Repeat brachial artery ultrasound imaging of the same subject after 1 hour using the same operator and vascular ultrasound equipment

SECONDARY OUTCOMES:
Incidence of emergent adverse device effects (ADEs) according to CTCAE v4.03 | 1 day
  Spontaneous ADEs reported by the subject and inquiry into emergence of expected/unexpected ADEs

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Lenehan, MD PhD, Study Chair — Everist Health
Locations (2):
- United States (2):
  - Yale University Prevention Research Center, Derby, Connecticut
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No